CLINICAL TRIAL: NCT06932341
Title: Use of a BPA to Promote High Value Care in Bronchiolitis: A Randomized Controlled Study
Brief Title: Leveraging Electronic Health Record Tools to Improve the Evidence-Based Treatment of Children Hospitalized With Bronchiolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00456658
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Bronchiolitis
Keywords: best practice advisory; clinical decision support; clinical guideline; clinical pathway
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No BPA (No Intervention): Clinicians will not be exposed to a BPA about the care of bronchiolitis. The participants will still have access to the EHR-embedded, evidence-based clinical guideline.
- Interruptive BPA (Experimental): Clinicians will be exposed to an interruptive BPA directing the clinician to reference the EHR-embedded, evidence-based clinical guideline for the care of bronchiolitis.
  Interventions: Other: Interruptive
- Non-interruptive BPA (Experimental): Clinicians will be exposed to an non-interruptive BPA directing the clinician to reference the EHR-embedded, evidence-based clinical guideline for the care of bronchiolitis.
  Interventions: Other: Non-interruptive

INTERVENTIONS:
Other: Non-interruptive — Non-interruptive BPA (appears as a visual cue but does not require clinicians to alter workflows) directing clinicians to reference the EHR-embedded, evidence-based clinical guideline for the care of bronchiolitis.
  Arms: Non-interruptive BPA
Other: Interruptive — Interruptive BPA (requires clinicians to interact with the alert to continue the workflow) directing clinicians to reference the EHR-embedded, evidence-based clinical guideline for the care of bronchiolitis.
  Arms: Interruptive BPA

SUMMARY:
The goal of this experimental study is to learn whether different types of best practice advisories (BPAs) that direct clinicians to reference clinical guidelines embedded in the electronic health record (EHR) increase the delivery of evidence-based care in children presenting to the hospital with bronchiolitis. The main questions it aims to answer are:

* Do BPAs improve clinicians' delivery of guideline-concordant care in bronchiolitis?
* Do interruptive BPAs improve guideline-concordant care of bronchiolitis more than non-interruptive BPAs?

Researchers will compare the treatment and outcomes of patients whose clinicians did not receive a BPA, to those whose clinicians received a non-interruptive BPA, to those whose clinicians received an interruptive BPA.

Patients will continue to receive standard hospital care for bronchiolitis.

Clinicians will:

* retain access to an EHR-embedded clinical guideline for bronchiolitis care
* be exposed to either no BPA, a non-interruptive BPA, or an interruptive BPA promoting the EHR-embedded clinical guideline (randomized per patient encounter)

DETAILED DESCRIPTION:
Bronchiolitis, a viral respiratory illness affecting infants and toddlers, is the most common reason children less than 2 years old are hospitalized. However, many children admitted with bronchiolitis receive unnecessary treatments that do not hasten recovery and may even cause harm. Despite evidence that the best treatment for bronchiolitis is supportive care (i.e. oxygen and hydration support), clinicians continue to overuse certain therapies, leading to longer hospital stays, higher costs, and increased stress for families.

The investigators will study the effects of BPAs, which are real-time alerts within the EHR. The BPAs in this study promote the use of an evidence-based care guideline for bronchiolitis that is embedded within the EHR. There are multiple BPA designs commonly used in EHRs: 1) interruptive BPAs, which require clinicians to interact with the alert to continue the clinician's workflow; and 2) non-interruptive BPAs, which appear as visual cues but do not require clinicians to alter workflows.

ELIGIBILITY:
Patient Inclusion Criteria:

* Children <=24 months of age presenting to the emergency room and/or hospitalized (under observation or inpatient status) with bronchiolitis at one of three study sites.

Patient Exclusion Criteria:

* Current encounter is birth-encounter
* Currently hospitalized in an ICU
* Hospitalized with length of stay >14 days

Clinician Inclusion Criteria:

* Physicians and advanced practice providers entering the patient's chart or orders entry activity for Emergency Department (ED) and inpatient encounters

Clinician Exclusion Criteria:

* Physicians and advanced practice providers who do not enter the patient's chart or orders entry activity

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Composite score of guideline-discordant care per hospital encounter | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
  Guideline-discordant care will be defined as a composite score incorporating number of chest X-rays, number of bronchodilator treatments, and numbers of hours spent on subtherapeutic rates of high-flow nasal cannula

SECONDARY OUTCOMES:
Hospital length of stay (hours) | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Duration of oxygen treatment (hours) | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Duration of high-flow nasal cannula treatment (hours) | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Number of Participants Transferred to intensive care unit | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Number of chest X-rays | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Number of bronchodilator treatments | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
Time spent on subtherapeutic rates of high-flow nasal cannula (hours) | From enrollment to the end of hospital stay, approximately 3 days
  Subtherapeutic rates of high-flow nasal cannula will be defined as <1 Liter/kilogram/minute
Number of Participants with Hospital readmission within 7 days | From enrollment to 7 days after hospital discharge

OTHER OUTCOMES:
Number of clinician interactions with clinical guideline | From enrollment to the end of ED encounter (approximately <24 hours) for non-hospitalized patients; End of hospital stay (approximately 2-4 days) for hospitalized patients
  To be measured based upon total number of interactions, as well as number of orders placed directly from clinical guideline interface

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bodnar, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No